CLINICAL TRIAL: NCT03057054
Title: The Effectiveness of Lactobacillus Plantarum (LBP, IND# 17339) in Preventing Acute Graft-Versus-Host Disease (GvHD) in Children Undergoing Alternative Hematopoietic Progenitor Cell Transplantation (HCT)
Brief Title: Lactobacillus Plantarum in Preventing Acute Graft Versus Host Disease in Children Undergoing Donor Stem Cell Transplant
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ACCL1633; NCI-2017-00208 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCL1633 (Other: Children's Oncology Group); COG-ACCL1633 (Other: DCP); ACCL1633 (Other: CTEP); R01CA201788 (NIH); UG1CA189955 (NIH)
Record Dates: First submitted 2017-02-15; First posted 2017-02-17 (Actual); Results first posted 2023-07-17 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Acute Graft Versus Host Disease; Hematopoietic and Lymphatic System Neoplasm; Leukemia; Lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma | interventions — Stem Cell Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (Lactobacillus plantarum, alloHCT) (Experimental): Patients receive Lactobacillus plantarum strains 299 and 299v PO or through NJ, NG or G tube QD on day 1 of transplant conditioning regimen to 56 days post alloHCT. Patients undergo alloHCT at day 0.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Biological: Lactobacillus plantarum strain 299; Biological: Lactobacillus plantarum strain 299v
- Arm II (placebo, alloHCT) (Placebo Comparator): Patients receive placebo PO or through NJ, NG or G tube QD on day 1 of transplant conditioning regimen to 56 days post alloHCT. Patients undergo alloHCT at day 0.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Other: Placebo Administration

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo alloHCT
  Other Names: Allogeneic; Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
Biological: Lactobacillus plantarum strain 299 — Given PO or via NJ, NG or G tube
  Other Names: DSM 6595; LACTOBACILLUS PLANTARUM 299
  Arms: Arm I (Lactobacillus plantarum, alloHCT)
Biological: Lactobacillus plantarum strain 299v — Given PO or via NJ, NG or G tube
  Other Names: DSM 9843; LACTIPLANTIBACILLUS PLANTARUM 299V; Lp 299v
  Arms: Arm I (Lactobacillus plantarum, alloHCT)
Other: Placebo Administration — Given PO or via NJ, NG or G tube
  Arms: Arm II (placebo, alloHCT)

SUMMARY:
This randomized phase III trial studies how well Lactobacillus plantarum works in preventing acute graft versus host disease in children undergoing donor stem cell transplant. Lactobacillus plantarum may help prevent the development of gastrointestinal graft versus host disease in children, adolescents, and young adults undergoing donor stem cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine efficacy of orally-administered Lactobacillus plantarum (LBP) in preventing the development of gastrointestinal (GI) acute graft versus host disease (aGvHD) in children and adolescents undergoing alternative donor allogeneic hematopoietic cell transplantation (alloHCT).

EXPLORATORY OBJECTIVES:

I. To determine whether orally-administered LBP decreases the incidence of grade II-IV aGvHD following alternative donor alloHCT.

II. To determine whether LBP administration maintains intestinal integrity as measured by mean serum citrulline levels and reduction in mucosal barrier injury (MBI) bacteremia.

III. To measure the effects of LBP on the intestinal flora phylogenetic composition during and after alternative donor alloHCT using 16S ribosomal ribonucleic acid (rRNA) gene deep sequencing.

IV. To measure effects of LBP on intestinal flora function during and after alternative donor alloHCT using metagenomic and metabolite profiling.

V. To measure proposed immunomodulatory effects of LBP in mean serum levels of alloreactive-induced inflammatory cytokines (IL-2, IL-6, IL-12p70, IFN gamma, TNF alpha, etc) in patients receiving LBP compared to placebo.

VI. To determine whether LBP administration reduces the incidence of Clostridium difficile-associated diarrhea in alternative donor HCT patients.

VII. To determine whether LBP administration reduces hospital days within the first 120 days post hematopoietic cell transplant (HCT).

VIII. To define the safety of orally administered LBP strains 299 and 299v in alternative donor HCT patients as measured by incidence of Lactobacillus plantarum bacteremia.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive Lactobacillus plantarum strains 299 and 299v orally (PO) or through nasojejunal (NJ), nasogastric (NG) or gastronomy (G) tube once daily (QD) on day 1 of transplant conditioning regimen to 56 days post alloHCT. Patients undergo alloHCT at day 0.

ARM II: Patients receive placebo PO or through NJ, NG or G tube QD on day 1 of transplant conditioning regimen to 56 days post alloHCT. Patients undergo alloHCT at day 0.

After completion of study treatment, patients are followed up for 120 days from alloHCT.

ELIGIBILITY:
Inclusion Criteria:

* All clinical and laboratory studies, if applicable, must be obtained within 21 days prior to start of protocol therapy (repeat if necessary); protocol therapy must begin within 6 months of study enrollment
* Patient must have a diagnosis that is managed with an alternative donor allogeneic hematopoietic cell transplant
* Patients must have a Lansky (for patients =< 16 years of age) or Karnofsky (for patients > 16 years of age) performance status score of >= 70; patients who are unable to walk because of a chronic underlying condition (such as paralysis), but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing performance score
* Hematopoietic cell transplant (HCT)

  * Patient must be receiving cells from alternative donor defined as one of the following:

    * Unrelated donor with a complete human leukocyte antigen (HLA) match or a 1 or 2 HLA mismatch, considering only HLA-A, HLA-B, HLA-C, and HLA-DRB1
    * Related donor with a 1 or more HLA mismatch (including haplo-identical)
    * Note: History of HCT or other cellular therapy (e.g. chimeric antigen receptor [CAR]-T cells, donor lymphocyte infusions) is permitted

Exclusion Criteria:

* Patient plans on receiving stem cells from a matched (8/8) related donor
* Patient has used a probiotic dietary supplement within the previous 30 days of enrollment; (consumption of yogurt products is allowed)
* Patient has a history of severe GI tract insult including but not limited to previous bowel perforation, grade 4 neutropenic colitis or typhlitis, inflammatory bowel syndrome, short small bowel syndrome (Crohn's disease, ulcerative colitis), history of gastrointestinal GVHD, or history of bowel resection
* Patient has a medical, psychiatric or social issue that would compromise patient safety or compliance with protocol therapy, or interfere with consent, study participation, follow up, or interpretation of study results
* Female patients who are pregnant are not eligible; women of childbearing potential require a negative pregnancy test prior to enrollment
* Patient has diarrhea at the time of enrollment which is Clostridium difficile toxin positive
* Patient is receiving antibiotic therapy for an active bacterial infection
* Patient is allergic to all third or fourth generation cephalosporins, carbapenems, and all aminoglycosides, which are used to empirically treat LBP bacteremia

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 173 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Nieder, Principal Investigator — Children's Oncology Group
Locations (43):
- United States (40):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Riley Hospital for Children, Indianapolis, Indiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - New York Medical College, Valhalla, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
- Canada (3):
  - Alberta Children's Hospital, Calgary, Alberta
  - Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment through day 120 post-stem cell infusion
Period: Overall Study
Arm/Group | Arm I (Lactobacillus Plantarum, alloHCT) | Arm II (Placebo, alloHCT)
Started | 85 | 88
Prior to Initial Stem Cell Infusion (Patients who started protocol therapy (either placebo or LBP, depending on randomization) after enrollment and prior to receiving their initial stem cell infusion.) | 83 | 86
Initial Stem Cell Infusion (Patients who received initial stem cell infusion within 6-months of study enrollment after initiating protocol therapy (LBP or placebo).) | 78 | 81
Completed | 74 | 80
Not Completed | 11 | 8
Not completed — Death | 4 | 4
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Ineligible | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Lactobacillus Plantarum, alloHCT) | Arm II (Placebo, alloHCT) | Total
Number analyzed (Participants) | 85 | 88 | 173
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 74 | 76 | 150
  Between 18 and 65 years | 11 | 12 | 23
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.7 (6.0) | 12.1 (5.6) | 11.4 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 35 | 64
  Male | 56 | 53 | 109
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 21 | 37
  Not Hispanic or Latino | 64 | 61 | 125
  Unknown or Not Reported | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 13 | 27
  White | 49 | 60 | 109
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 15 | 11 | 26
Region of Enrollment [Number; unit: participants]
  United States | 78 | 83 | 161
  Canada | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Stage 1-4 Gastrointestinal (GI) Acute Graft Versus Host Disease (aGVHD)
Description: The proportion of eligible patients having stage 1-4 GI aGvHD occur from Day 0 through Day 120 will be compared between the two arms.
Time Frame: Up to 120 days post stem cell infusion
Population: 2 patients were excluded because they were not eligible (1 patient from Group 1 and 1 patient from Group 2). 2 patients were excluded because they did not initiate treatment (1 patient from Group 1 and 1 patient from Group 2). 10 patients were excluded because they never received a stem cell infusion within 6 months of enrollment (5 patients from Group 1 and 5 patients from Group 2).
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Arm I (Lactobacillus Plantarum, alloHCT) | Arm II (Placebo, alloHCT)
Number analyzed (Participants) | 78 | 81
Proportion of patients | 0.15 [0.08 to 0.25] | 0.15 [0.08 to 0.24]

2. Other Pre Specified Outcome: Incidence of Grade II-IV Overall Graft Versus Host Disease
Description: A similar analysis approach will be used as described for the primary outcome measure but using the dichotomous cumulative incidence of grade II-IV acute graft versus host disease as the endpoint measure.
Time Frame: Up to 120 days post stem cell infusion
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Incidence of Blood Stream Infection
Description: The risk of mucosal barrier blood stream infections will be compared between two groups.
Time Frame: Up to 120 days post stem cell infusion
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Incidence of Clostridium Difficile (C. Diff)-Associated Diarrhea
Description: Proportion of C. diff-associated diarrhea during the study period will be compared between arms.
Time Frame: Up to 120 days post stem cell infusion
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Serum Levels of Citrulline
Description: The change in citrulline levels from baseline to each of the time points (days 7, 14, 28, 56, and 120 post-infusion) will be summarized and described by arm.
Time Frame: Up to 120 days post stem cell infusion
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Bacterial Genes and Pathways, and Bacterial Metabolites (Blood/Stool Measures of Intestinal Flora - Function and Phylogenetic Composition)
Description: LBP introduction on the intestinal flora via LBP administration will be compared with bacterial genes and pathways, and bacterial metabolites via correlation analyses. Also, dDescriptive analysis will be used to examine the association between the graft versus host disease outcomes (GI aGvHD and overall GvHD) and bacterial genes, pathways, and metabolites.
Time Frame: Up to 120 days post stem cell infusion
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Blood/Stool Measures of Intestinal Flora Assessed Using Sequencing
Description: The association between Lactobacillus plantarum administration and bacterial genes and pathways, and bacterial metabolites will be evaluated.
Time Frame: Up to 120 days post stem cell infusion
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Levels of Pro-inflammatory Cytokines
Description: The effects of Lactobacillus plantarum on pro-inflammatory (LBP) cytokines in allogeneic hematopoietic cell transplantation recipients will be examined by comparing levels across arms.
Time Frame: Up to 120 days post stem cell infusion
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Hospital Days
Description: Total hospital days over the study period is calculated as the duration between the date of admission for conditional therapy and the date of discharge (or the study end date). Hospital days will be compared between arms.
Time Frame: Up to 120 days post stem cell infusion
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Incidence of Lactobacillus Plantarum Bacteremia
Description: Patients who have at least one incidence (positive) of lactobacillus plantarum during any reporting period is considered evaluable for this aim. The proportion of patients experiencing lactobacillus plantarum bacteremia during the study period will be compared between arms.
Time Frame: Up to 120 days post stem cell infusion
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Collected Adverse Events within the 100 day observation period
Description: Adverse event reporting is collected routinely using case report forms. SAE field contains NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted via expedited reporting (NCI AdEERs / CAeRs). The AE field contains grade 3 and higher CTCAEs reported on study excluding those that were reported as SAEs. All-Cause Mortality events were monitored/assessed in all randomized participants. Serious and Other Adverse Events were monitored/assessed only in the eligible participants.
Arm/Group | Arm I (Lactobacillus Plantarum, alloHCT) | Arm II (Placebo, alloHCT)
All-Cause Mortality (participants affected / at risk) | 4/85 | 4/88
Serious Adverse Events (participants affected / at risk) | 5/84 | 8/87
Other Adverse Events (participants affected / at risk) | 9/84 | 9/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Lactobacillus Plantarum, alloHCT) (N=84) | Arm II (Placebo, alloHCT) (N=87)
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Bacteremia (Infections and infestations) | 1 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 1
Cytomegalovirus infection reactivation (Infections and infestations) | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Death NOS (General disorders) | 1 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 1
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 1 | 0
Hepatic hemorrhage (Hepatobiliary disorders) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 2 | 4
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sinusoidal obstruction syndrome (Hepatobiliary disorders) | 2 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0
Typhlitis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Viremia (Infections and infestations) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Lactobacillus Plantarum, alloHCT) (N=84) | Arm II (Placebo, alloHCT) (N=87)
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Anemia (Blood and lymphatic system disorders) | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Autoimmune disorder (Immune system disorders) | 1 | 0
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 2 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Infections and infestations - Other, specify (Infections and infestations) | 2 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 1 | 1
Sinusoidal obstruction syndrome (Hepatobiliary disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Cytomegalovirus (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/54/NCT03057054/Prot_SAP_000.pdf